CLINICAL TRIAL: NCT01171209
Title: REsPonse to Interferon-Alpha in InterfeRon-β Neutralizing Antibody Positive Multiple Sclerosis Patients
Acronym: REPAIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinda Magyari (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Melinda Magyari, M.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-016824-29; 2009-016824-29 (EudraCT Number)
Record Dates: First submitted 2010-07-08; First posted 2010-07-28 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon-beta; Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IFN-alfa (Experimental): One single injection of human leukocyte IFN-α (Multiferon® ) 6 MIU s.c.
  Interventions: Drug: Interferon-beta and human leukocyte Interferon-α
- Interferon-beta (Experimental): One single injection of IFN-beta followed by blood test for MxA9.12 hours after injection
  Interventions: Drug: Interferon-beta and human leukocyte Interferon-α

INTERVENTIONS:
Drug: Interferon-beta and human leukocyte Interferon-α — One single injection of interferon(IFN)- β and one single injection of human leukocyte IFN-α (Multiferon® ) 6 MIU s.c. with 1-7 days follow-up.
  Other Names: IFN-beta : Rebif, Betaferon; IFN-alfa: Multiferon®

SUMMARY:
The purpose of the study is to determine if Interferon-alfa is effective and safe in multiple sclerosis patients who developed neutralizing antibodies for Interferon-beta.

DETAILED DESCRIPTION:
Patient with NAbs developed during IFN-β therapy do not have any longer beneficial effect of any IFN-β preparation and IFN-β has to be replaced with another therapy that may be less effective or carry along serious adverse effects. Hence, many NAb positive patients wish to continue IFN therapy, and these patients might benefit from treatment with IFN-α as both IFN-α and IFN-β are type I interferons that bind to the same interferon receptor (IFNAR). A full in vivo response to human IFN-α (Multiferon) comparable to that seen after IFN-β induction would suggest that the same therapeutic effect could be obtained with human IFN-α (Multiferon).We measure in vivo response of MxA 9-12 hours after administration of human IFN-α (Multiferon) and four other known IFN response markers measured with rt-PCR.

As controls, NAb negative MS patients with a full in vivo MxA response will be studied.

ELIGIBILITY:
Inclusion Criteria:

* The subject must give written informed consent prior to any study related activities
* Subject age must be between 18 and 55 (both included)
* The subject must have MS according to McDonald criteria
* The subject must have disability equivalent to EDSS of 5.5 or less
* The subject must have been treated with any IFN-β preparation for at least 12 months at any time
* The subject must have been shown to be NAb positive and without no in vivo mRNA MxA response within the last 12 months
* The subject must be prepared and considered able to follow the protocol

Exclusion Criteria:

* The subject must not have conditions that might give rise to similar symptoms as MS
* The subject must not have received any immunomodulatory or immunosuppressive treatment (other than IFN-β or glatiramer acetate) 6 months prior to the screening visit
* The subject must not have received mitoxantrone, cyclophosphamide, treosulphane, natalizumab, daclizumab, rituximab, alemtuzumab, cladribine, or any experimental therapy at any time
* The subject must not have undergone previous total body irradiation, total lymphoid irradiation, stem cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
* The subject must not have received treatment with glucocorticoids or ATCH later than 2 month prior to the screening visit
* The subject must not have alcohol and drug dependency
* The subject must not have cardiac or renal insufficiency
* The subject must not have any systemic disease that can influence the subject's safety or compliance
* Subjects may be male or female. Women of child-bearing potential must be sexually inactive or practice a medically acceptable method of birth control. Acceptable methods include oral contraceptive, contraceptive patch, long-acting injectable contraceptive, or double-barrier method (condom or IUD with spermicide)
* The subject must not have known or suspected allergy to IFN-α
* The subject must not have participated in any other study within 3 months prior to the screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
In vivo mRNA MxA response | 9-12 hours after injection of one dose Interferon-alfa
  The primary objective of this study is to compare the in vivo mRNA MxA response to IFN-α with the in vivo mRNA MxA response to IFN-β

SECONDARY OUTCOMES:
Determining response marker: IL10 | 9-12 hours after adminstration of Interferon-alfa
  The in vivo response to IFN-α of known IFN response marker: interleukin-10 (IL10),
Determining response marker:TRAIL | 9-12 hours after administration of IFN-alfa
  Determining tumor necrosis factor-related apoptosis-inducing ligand (TRAIL)
Determining response marker IFI27 | 9-12 timer after administration of IFN-alfa
  Determining IFN-α-inducible protein 27 (IFI27),
Determining response marker:CXCL10 at mRNA level | 9-12 hours after IFN-alfa administration
  Determining :Chemokine CXCL10 at mRNA level
Changes i Neutralizing antibodies Nabs | 9-12 hours after administration of IFN-alfa
  Measuring changes in Neutralising antibodies 9-12 hours after treatment with one dose IFN-alfa

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Magyari, M.D., Principal Investigator — Danish Multiple Sclerosis Research Center

REFERENCES:
- [Derived] Magyari M, Bach Sondergaard H, Sellebjerg F, Soelberg Sorensen P. Preserved in vivo response to interferon-alpha in multiple sclerosis patients with neutralising antibodies against interferon-beta (REPAIR study). Mult Scler Relat Disord. 2013 Apr;2(2):141-6. doi: 10.1016/j.msard.2012.10.001. Epub 2012 Dec 11. PMID 25877635